CLINICAL TRIAL: NCT06568354
Title: The Effects of Yoga and Motor Control Exercises on Pain Perception, Function, and Pain Cognition in Patients With Chronic Neck Pain
Brief Title: The Effects of Yoga and Motor Control Exercises in Patients With Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Prof, Spine Health Unit, Principal Investigator, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTREK24/24
Record Dates: First submitted 2024-08-16; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Chronic Neck Pain
Keywords: neck pain; exercise; cognition; yoga; motor control; function
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Active Comparator): A yoga exercise program will be applied in two sessions per week, a total of eight weeks.
  Interventions: Other: Yoga
- Motor Control Exercise Group (Active Comparator): Motor control exercise program will be applied two sessions per week, totally eight week.
  Interventions: Other: Motor control exercises

INTERVENTIONS:
Other: Yoga — The yoga program was applied to all patients in this group, accompanied by a physiotherapist. Sessions included selected breathing, warm-up, and relaxation exercises.
  Arms: Yoga Group
Other: Motor control exercises — Motor control exercises with three different progressive phases were applied to all patients in this group accompanied by a physiotherapist.
  Arms: Motor Control Exercise Group

SUMMARY:
Identification of the effects of yoga and motor control exercises on pain intensity, pain sensitivity, function, and pain cognition in individuals with neck pain.

DETAILED DESCRIPTION:
Patients participating in the study were divided into two parallel groups. The patients in the motor control exercise group were instructed to perform motor control exercises, which consist of strengthening of the deep cervical flexors, deep cervical extensors, and axioscapular muscles; stretching exercises; postural correction exercises, and patients in the yoga group were instructed to perform a yoga program, which consists of breathing, relaxation, and flexibility exercises.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain
* Must be pain at least 3 months

Exclusion Criteria:

* History of any cervical spine surgery
* Presence of neurological deficit
* Having been diagnosed with cardiovascular or systemic diseases that would prevent him/her from taking exercise training.
* Inflammatory, infectious, or tumoral disease of the vertebra
* Severe/progressive scoliosis, spinal stenosis, spondylolisthesis
* had been diagnosed with a neurological disease
* were currently pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in Functional Disability | Change from baseline in functional status at 8 weeks
  The Neck Disability Index, modified from the Oswestry Low Back Pain Questionnaire and adapted to the cervical region by Vernon et al. in 1991, will be used to assess disability due to neck pain. In the neck disability index, a score of 0-4 is defined as no disability, a score of 5-14 is defined as mild disability, a score of 15-24 is defined as moderate disability, a score of 25-43 is defined as severe disability and a score above 35 is defined as total disability.

SECONDARY OUTCOMES:
Changes in Pain Intensity | Change from baseline in pain intensity at 8 weeks
  It will be evaluated with the Numeric Pain Scale. Individuals will be told that '0' means the absence of pain and '10' means the presence of unbearable pain, they will be asked to indicate the average and maximum pain intensity they have experienced in the last 48 hours and the average pain intensity in the last week between 0-10 and their responses will be recorded.
Changes in Pain Sensitivity | Change from baseline in pain sensitivity at 8 weeks
  Pressure pain threshold (PPT) assessment will be performed with a device called algometer to evaluate the individuals' pain sensitivity. Initially, 2 trials are performed on the extensor muscles of the forearm to familiarize the participant with the procedure. Afterwards, the person is positioned according to the area to be measured and the measurement points are marked with a pencil. The algometer is placed perpendicular to the skin and a constant pressure is applied. The participant is asked to say "stop" when the feeling of pressure or discomfort turns into a clear sensation of pain. Three measurements are taken at 30 s intervals at each site. The values are averaged and recorded. In this study, right/left C1-C2 and C5-6 articular region, upper part of the Trapezius muscle, Deltoid muscle insertion, lateral epicondyle will be used as measurement points. Measurements will also be made on the Tibialis anterior muscle to assess overall pain sensitivity.
Changes in Alexithymia | Change from baseline in alexithymia at 8 weeks
  The alexithymia will be assessed by the Toronto Alexithymia Scale (TAS). The scale is a Likert-type self-assessment scale consisting of 20 items and scored between 1-5. Difficulties in recognizing emotions (TAS-1), difficulty in speaking emotions (TAS-2), extroverted thinking (TAS-3) subscales. The individual is asked to select the best option for each item from "Never", "Rarely", "Sometimes", "Often" and "Always". The higher the score, the higher the level of alexithymia.
Changes in Cognitive Function | Change from baseline in cognitive function at 8 weeks
  The Montreal Cognitive Assessment Questionnaire (MoCA) will be used to assess the cognitive function of individuals. MoCA was developed as a rapid screening test for mild cognitive impairment. MoCA assesses various cognitive functions such as attention and concentration, creative functions, memory, language, visual structuring skills, abstract thinking, computation, and orientation. The application of MoCA takes about 10 minutes. The maximum total score of the test is 30. A score of 21 or above is considered normal.
Changes in Pain Catastrophizing | Change from baseline in pain catastrophizing at 8 weeks]
  The Pain Catastrophizing Scale will be used to evaluate the individual's pain-related catastrophizing thoughts. In the scale consisting of thirteen questions, each question is scored between 0-4. It is graded as "0" never, "1" mildly, "2" moderately, "3 severely, "4" always. The answers to the thirteen questions are summed to obtain a score.
Changes in Kinesiophobia | Change from baseline in kinesiophobia at 8 weeks
  The Tampa Kinesiophobia Scale (TKS) will be used to assess the kinesiophobia levels of individuals. The TKS is a 17-question Likert scale that examines activity-related injury/reinjury and fear-avoidance parameters. The score on the scale ranges from 17-68, and the higher the score, the higher the level of kinesiophobia.
Changes in Neck Awareness | Change from baseline in neck awareness at 8 weeks]
  The Fremantle Neck Awareness Questionnaire will be used to assess how individuals perceive the neck area relative to their body. In the questionnaire, there are 9 questions measuring how individuals perceive their neck relative to their body and how they perceive their body position, and the questions are answered in Likert type as "0" I never feel like this, "4" always or often feel like this.
Changes in Body Awareness | Change from baseline in body awareness at 8 weeks
  The Body Awareness Rating Questionnaire will be used to assess the body awareness of individuals. This self-reported questionnaire consists of 4 different factors indicating different aspects of body awareness. The factors assess body awareness in terms of function, feeling/emotion, mood and awareness. Each item is scored on a 7-point Likert-type scale. Scores for each factor range from 6 to 42, with higher scores indicating greater body awareness
Changes in Central Sensitization | Change from baseline in central sensitization at 8 weeks
  The Central Sensitization Scale will be used to assess central sensitization. The Central Sensitization Scale is a valid and reliable scale that identifies whether patients' existing symptoms are associated with central sensitization. It consists of two parts. Part A consists of 25 items, including somatic and emotional symptoms related to central sensitization, while part B inquires about previous diagnoses of central sensitization syndromes or related diseases. The frequency of symptoms is assessed on a four-point Likert scale from 0 (never) to 4 (always). The total score ranges from 0 to 100, with higher scores indicating a high degree of central sensitization.
Changes in Hand Grip Strength | Change from baseline in hand grip strength at 8 weeks
  A Hydraulic Hand Dynamometer will be used to measure hand grip strength. The assessment will be performed using the standard measurement method of the American Association of Hand Therapists. For the assessment, the participant is held in an upright sitting position, feet in contact with the floor, arm next to the body, elbow in 90◦ flexion, forearm and wrist in a neutral position. To assess hand grip strength, the evaluated participant's hand is placed so that it grasps the second measurement range of the dynamometer. Grip strength will be assessed by changing hands between measurements and three measurements will be taken for each hand. An interval of 15 seconds will be used between each measurement. The average of the three measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Ulger, Prof, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho WS, Park CB, Kim BG. Effects of exercise therapy on pain and disability in patients with non-specific neck pain: A systematic review and meta-analysis. J Bodyw Mov Ther. 2023 Oct;36:213-220. doi: 10.1016/j.jbmt.2023.07.010. Epub 2023 Jul 13. PMID 37949563
- [Background] Cramer H, Klose P, Brinkhaus B, Michalsen A, Dobos G. Effects of yoga on chronic neck pain: a systematic review and meta-analysis. Clin Rehabil. 2017 Nov;31(11):1457-1465. doi: 10.1177/0269215517698735. Epub 2017 Mar 9. PMID 29050510
- [Background] Akodu AK, Nwanne CA, Fapojuwo OA. Efficacy of neck stabilization and Pilates exercises on pain, sleep disturbance and kinesiophobia in patients with non-specific chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:411-419. doi: 10.1016/j.jbmt.2020.09.008. Epub 2020 Oct 3. PMID 33992276
- [Background] Rasmussen-Barr E, Halvorsen M, Bohman T, Bostrom C, Dedering A, Kuster RP, Olsson CB, Rovner G, Tseli E, Nilsson-Wikmar L, Grooten WJA. Summarizing the effects of different exercise types in chronic neck pain - a systematic review and meta-analysis of systematic reviews. BMC Musculoskelet Disord. 2023 Oct 12;24(1):806. doi: 10.1186/s12891-023-06930-9. PMID 37828488